CLINICAL TRIAL: NCT03568019
Title: PET Avidity in Cachexia-Inducing Lung and Gastrointestinal Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Anne Gilmore, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 092013-001
Record Dates: First submitted 2018-05-14; First posted 2018-06-26 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Cachexia; Cancer
MeSH Terms: conditions — Cachexia; Neoplasms | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Retrospective study — No subjects will be contacted or recruited. All data will be acquired retrospectively.

SUMMARY:
PET has an established role in the initial staging of patients with newly diagnosed lung and gastrointestinal tumors.PET avidity is described with both maximum and mean standardized uptake values.Malignant cells have increased activity on PET, defined as the standardized uptake value (SUV), with increased uptake of FDG in tumor due to elevated levels of GLUT receptors, elevated intracellular levels of hexokinase and increased rates of glycolysis. However, there is a subset of patients with lung and gastrointestinal tumors that are not PET avid.These patients may present with clinically and systemically aggressive disease with a declining performance status and/or weight loss.

DETAILED DESCRIPTION:
This study will be a retrospective review of patients in the tumor registry with lung and gastrointestinal tumors, not limited to but including small and non-small cell lung cancers, stomach cancer, small intestinal cancer, colon cancer, rectal cancer, liver and intrahepatic bile duct cancers, gallbladder and extrahepatic bile duct cancers, and pancreatic cancer.

There will be a maximum of 10,000 charts/records that will be reviewed to compile the data. Data to be collected will include patients' name, medical record number, date of birth, race, ethnicity, gender, medical history, medications, vital and performance status, vital signs including weight and body mass index, date of cancer diagnosis, clinical and pathologic stage, pathology, treatment course, prior treatment, location of primary lesion, and smoking history. CT and PET findings to be reviewed include the number of involved lymph nodes, size of primary tumor, average/maximum PET avidity in both the primary tumor and involved lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically proven lung and gastrointestinal cancers, stages I-IV with PET and/or CT within 6 weeks of diagnosis.

Exclusion Criteria:

There will be no absolute exclusion criteria as long as the inclusion criteria have been met.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically proven lung and gastrointestinal cancers
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
A retrospective review to determine if PET can be used to identify cachexia-inducing lung and gastrointestinal tumors | 10 years
  The goal of this assessment is to identify patients with lung and gastrointestinal tumors and collect the data on tumor stage location, histology, PET avidity, and weight loss/performance status so that it will be possible to correlate SUV values associated with cachexia by using CTCAE version 4.0 to collect and log AE and SAE related to cachexia.

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Gilmore, MD, Principal Investigator — UTSW School of Health Professions - Clinical Nutrition Admin; Orhan Oz, MS, Principal Investigator — UTSW Radiation Oncology
Locations (1):
- UT Southwestern Medical Centre, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided